CLINICAL TRIAL: NCT02206490
Title: Trial of Naltrexone and Dextromethorphan for Gulf War Veterans Illnesses
Brief Title: Trial of Naltrexone and Dextromethorphan for Gulf War Illness
Acronym: GWI Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, William J. Meggs, Professor, East Carolina University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 090562
Record Dates: First submitted 2012-08-24; First posted 2014-08-01 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Gulf War Illness
Keywords: Gulf War Illness; treatment; dextromethorphan; naltrexone
MeSH Terms: interventions — Naltrexone; Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Naltrexone Study Drug (Active Comparator): Subjects will take naltrexone 4.5 mg daily for three months.
  Interventions: Drug: naltrexone
- Naltrexone placebo (Placebo Comparator): Subjects will take a 3 month course of a placebo pill identical in appearance to the naltrexone study drug.
  Interventions: Drug: naltrexone
- dextromethrophan study drug (Active Comparator): subjects will take a sustained release dextromethorphan pill twice a day.
  Interventions: Drug: Dextromethorphan
- dextromethoprhan placebo (Placebo Comparator): Subjects will take a 3 month course of a placebo pill identical in appearance to the dextromethorphan study drug.
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Drug: naltrexone — Randomized controlled trial of naltrexone for Gulf War Illness.
  Arms: Naltrexone Study Drug; Naltrexone placebo
Drug: Dextromethorphan — Randomized controlled trial of dextromethorphan for Gulf War Illness
  Arms: dextromethoprhan placebo; dextromethrophan study drug

SUMMARY:
Veterans of the 1991 Gulf War who developed Gulf War Illness are being studied. Treatments with FDA approved generic drugs are being administered to see if they help with the symptoms of Gulf War Illness, such as chronic fatigue; difficulty with memory, concentration, and thinking; widespread chronic pain; and autonimic dysfunction. Drugs to be tested are dextromethorphan and naltrexone.

DETAILED DESCRIPTION:
Gulf war veterans' illnesses comprise distinct clusters of symptom-defined illnesses for which there are neither diagnostic tests nor effective treatments. Gulf war veterans had variable exposures to a number of chemicals, including organophosphate insecticides, pyrethrum-related insecticides, DEET, Pyridostigmine bromide, smoke from oil well fires, and Sarin gas. Gulf war veterans' illnesses may reflect an inflammatory cycle involving the brain which may be a common mechanism of many neurological conditions, whether initiated by toxic exposures, infection, or trauma. In this theory, central nervous system inflammation initiated by toxic exposures and sometimes exacerbated by subsequent exposures is a component of illness hypothesized to explain the neurological manifestations. Substance P release at sensory nerve endings is an explanation for the peripheral pain manifestations of illness.

This theory suggests that novel anti-inflammatory drugs may be of benefit in symptom-defined illnesses related to a cycle of inflammation. Dr. J. S. Hong's laboratory at the National Institute of Environmental Health Sciences has demonstrated that Morphine-related analogs, including Naltrexone and Dextromethorphan, have great potency in anti-inflammation and neuroprotective effects. Naltrexone is a safe and readily available generic medication. Dextromethorphan is also a safe and readily available generic medication that is available without a prescription as a cough medication. Results from several clinical trials showed that Naltrexone is effective in several inflammation-related diseases, such as neurogenic pain, movement disorders, etc. In addition, there were no obvious side effects in patients taking this drug for six months. This project will conduct randomized double-blinded studies for treating ill Gulf war veterans with Naltrexone and Dextromethorphan. Laboratory tests for markers of inflammation including neurogenic inflammation will be performed pre- and post-treatment, to see if these markers are elevated and if so, to see if treatment modulates these markers.

Ill Gulf veterans will be recruited through the media, veterans groups, and individual veteran activists. A screening telephone interview will be performed to determine if the veterans meet a modified Kansas case definition for inclusion. Those veterans who meet study criteria will be invited to participate. Eligible veterans will be invited for an initial visit that will consist of obtaining written informed consent, a medical history, physical examination, and laboratory testing. Institutional review board approval of the study will be in place. The pharmacy staff at the institution will prepare the medications and placebo in identical capsules.

ELIGIBILITY:
Inclusion Criteria:

* Served in the Gulf War and developed the symptoms of Gulf War Illness as described by the modified Kansas Case Definition

Exclusion Criteria:

* Pregnant women, nursing mothers, individuals requiring medications that have drug interactions with dextromethorphan or naltrexone, cancer not in remission, chronic infectious disease, liver disease, lupus, multiple sclerosis, stroke, under current treatment for schizophrenia, bipolar disorder/manic depression, and depression.
* Those with a history of current illicit drug use will be excluded. Individuals who have had recent surgery will not be enrolled until they have completely recovered from the surgery.
* Subjects participating in other clinical trials will be excluded.
* Those enrolled recently in a clinical trial will be enrolled after a washout period of one month.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Symptoms Scores | 28 weeks approximately
  Symptoms of Gulf War Illness will be scored by participants using a ten center meter scale.
  Scores will be collected at the end of 12 weeks/16 weeks/28weeks

SECONDARY OUTCOMES:
SF-36 | 28 weeks approximately
  Subjects will complete a standard health assessment tool, the SF-36, at the end of each course of therapy.
  Scores will be collected at 12 weeks/16 weeks/28 weeks
Connors Continuous Performance Test | 28 weeks approximately
  Subjects will take the Connors Continuous Performance Test at the end of each course of study drug or placebo.
  Scores will be collected at 12 weeks/16 weeks/28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Brody School of Medicine a East Carolina Univesity, Greenville, North Carolina, United States